CLINICAL TRIAL: NCT04968041
Title: Feasibility Trial Assessing Adherence and Response to a Ketogenic Dietary Intervention for Individuals at High Risk for Alzheimer's Disease
Brief Title: KNA Proof-of-Concept
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Julia Sheffler, Assistant Professor, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000111
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-08

CONDITIONS: Adherence, Treatment; Retention; Cognitive Impairment, Mild
MeSH Terms: conditions — Treatment Adherence and Compliance; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MI-CBT KNA Program (Experimental): 6-week group intervention using MI and CBT strategies to promote adherence to a ketogenic nutrition program.
  Interventions: Behavioral: Motivational Interviewing-Cognitive Behavioral Therapy Ketogenic Nutrition Adherence Program

INTERVENTIONS:
Behavioral: Motivational Interviewing-Cognitive Behavioral Therapy Ketogenic Nutrition Adherence Program — The intervention using strategies from motivational interviewing and cognitive behavioral therapy to promote motivation and adherence to ketogenic nutrition in older adults at high risk for Alzheimer's disease. The program is a 6-week, group program led by a psychologist and nutrition expert.
  Other Names: MI-CBT KNA Program

SUMMARY:
The intervention program proof-of-concept was assessed as a single-arm, within-subjects clinical study with a target enrollment of 10 participants with possible or probable amnestic MCI. The protocol required participants to complete a pre-intervention assessment within two weeks of beginning the intervention, attend seven, one-hour intervention group sessions across six weeks, complete a post-assessment and interview in the final week of the intervention, and complete weekly surveys throughout the intervention.

DETAILED DESCRIPTION:
The primary goal of the proof-of-concept phase is to use pre-post comparisons to determine if the treatment package can produce clinically significant improvements. Thus, our goal was to assess whether the MI-CBT KNA program influenced adherence to KN and cognitive outcomes. Of note, recruitment for the trial occurred in the weeks leading up to the COVID-19 pandemic, which substantially altered the original intervention and assessment design due to restrictions on in-person human subject research. While the original protocol included in-person assessments and group meetings, collection of multiple biological samples (i.e., lipid panels, basic vitals, inflammatory biomarkers), and weekly health assessments, these in-person components were modified or removed for completion during the COVID-19 pandemic. Pre-assessment and screening appointments described below were completed in-person prior to the COVID-19 pandemic. Thus, we completed pre-intervention neuropsychological assessments with participants at baseline prior to beginning the trial; however, immediately following baseline assessments, we fully revised the protocol to include only online, video, and phone contact. We moved the KNA program to an online platform (HIPAA-compliant Zoom), and assessments were changed to online surveys and video assessments. Individual testing of the video platform was completed prior to the trial, which successfully reduced technical problems.

The MI-CBT KNA Program proof-of-concept was assessed as a single-arm, within-subjects clinical study with a target enrollment of 10 participants with possible or probable amnestic MCI. The protocol required participants to complete a pre-intervention assessment within two weeks of beginning the intervention, attend seven, one-hour intervention group sessions across six weeks, complete a post-assessment and interview in the final week of the intervention, and complete weekly surveys throughout the intervention. Participants were mailed materials, including the participant workbook and food, macronutrient, and ketone logs. Participants were also sent two bottles of ketone urine test strips for daily testing and materials to complete follow-up assessments. Throughout the program, participants were instructed to titrate into full ketosis across the first four weeks of the program by gradually reducing total carbohydrate intake and increasing healthy fat intake (e.g., fish, nuts, avocado, olive oils etc.). Thus, participants were not expected to attain measurable ketone levels until the final weeks of the program.

ELIGIBILITY:
Inclusion Criteria:

* Final inclusion criteria included individuals who met criteria for "possible" Mild cognitive impairment (MCI), which was defined as the following: evidence of either subjective decline in memory and greater self-reported use of compensatory strategies OR poorer performance than expected in one or more cognitive domain OR limited evidence of impairment in both subjective and objective findings.

Exclusion Criteria:

* Presence of severe and/or unstable medical conditions
* diagnosable major neurocognitive disorder

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sheffler JL, Arjmandi B, Quinn J, Hajcak G, Vied C, Akhavan N, Naar S. Feasibility of an MI-CBT ketogenic adherence program for older adults with mild cognitive impairment. Pilot Feasibility Stud. 2022 Jan 22;8(1):16. doi: 10.1186/s40814-022-00970-z. PMID 35065656

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MI-CBT KNA Program
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | MI-CBT KNA Program
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.44 (3.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 5
  Black | 2
  Latino/Hispanic | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Repeatable Battery for Assessment of Neuropsychological Status (RBANS-Update) [Mean (Standard Deviation); unit: units on a scale] — Repeatable Battery for Assessment of Neuropsychological Status (RBANS-Update) Total Scaled Score. Scores are normed based on age, and 100 is considered average (50th percentile). Higher scores are associated with better cognitive functioning.
  units on a scale | 89.78 (9.135)
Adherence [Mean (Standard Deviation); unit: units on a scale] — Participants self-rated their adherence to the diet on a 1-10 scale, with higher scores corresponding to better adherence.
  units on a scale | 8.56 (1.87)

OUTCOME MEASURES:

1. Primary Outcome: Ketogenic Adherence
Description: Assessed based on reported ketone levels during the program (reporting at least one day or greater with trace amounts of ketones) using urinalysis ketone test strips administered at home by participants.
Time Frame: 6-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MI-CBT KNA Program
Number analyzed (Participants) | 9
Participants | 8

2. Primary Outcome: Acceptability
Description: Assessed based on qualitative feedback and online surveys described here: https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-022-00970-z.
  Participants also rated how well they felt the program helped them achieve their health-related goals 0 (none) to 3 (all).
Time Frame: 6-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MI-CBT KNA Program
Number analyzed (Participants) | 9
Participants
  All goals | 3
  Most | 1
  Some | 5

3. Primary Outcome: Retention
Description: Assessed based on attendance and % of participants who remained in the program from start to finish
Time Frame: baseline to 6-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MI-CBT KNA Program
Number analyzed (Participants) | 9
Participants | 9

4. Secondary Outcome: Cognitive Functioning
Description: Assessed using the total scaled score (age-normed) of the Repeatable Battery for the Assessment of Neuropsychological Status - Update. A score of 100 is considered "average" (50th percentile), and higher scores are considered better cognitive functioning. The outcome reported is the actual value at 6-weeks, rather than a change score.
Time Frame: Baseline and 6-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MI-CBT KNA Program
Number analyzed (Participants) | 9
score on a scale | 97.11 (11.14)

ADVERSE EVENTS:
Time Frame: Baseline to 3 months post-intervention (approximately 6 months)
Arm/Group | MI-CBT KNA Program
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT04968041/Prot_SAP_000.pdf